CLINICAL TRIAL: NCT01366300
Title: Estimation of the Effect of Intravenous Lidocaine on BIS-guided Propofol Requirements During General Anesthesia
Brief Title: Effect of Intravenous Lidocaine on BIS-guided Propofol Requirements During General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Fernando Altermatt, Pontificia Universidad Católica de Chile - Departamento de Anestesiología
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LPBIS-UC-2010
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-03

CONDITIONS: Intravenous Anesthetic Interaction "Unrecognized Condition"
MeSH Terms: interventions — Propofol; Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous lidocaine infusion (Active Comparator): Intravenous lidocaine infusion during total intravenous anesthesia with propofol administered by target controlled infusion
  Interventions: Drug: Intravenous lidocaine infusion; Drug: Propofol 1% (intravenous infusion); Procedure: Placement of arterial line
- Intravenous 0.9% saline infusion (Placebo Comparator): Intravenous 0.9% saline infusion during total intravenous anesthesia with propofol administered by target controlled infusion
  Interventions: Other: Placebo (0.9% saline infusion); Drug: Propofol 1% (intravenous infusion); Procedure: Placement of arterial line

INTERVENTIONS:
Drug: Intravenous lidocaine infusion — Once the dose of propofol required for general anesthesia is stabilized for 5 minutes with BIS values between 40 and 50, lidocaine 1% infusion is begun in a bolus of 1.5mg/kg for 5 minutes and then infused at 2 mg/kg/hr until the end of surgery (last skin suture is made).
  Arms: Intravenous lidocaine infusion
Other: Placebo (0.9% saline infusion) — Once the dose of propofol required for general anesthesia is stabilized for 5 minutes with BIS values between 40 and 50, 0.9% saline infusion is begun in a bolus of 1.5mg/kg for 5 minutes and then infused at 2 mg/kg/hr until the end of surgery (last skin suture is made).
  Arms: Intravenous 0.9% saline infusion
Drug: Propofol 1% (intravenous infusion) — Propofol is administered according to a widely-accepted pharmacokinetic model, initially dosed to a target controlled infusion (TCI) of 4.5 micrograms/ml, and titrated by step increases of 0.5 every minute until loss of conscience is obtained and BIS values are less than 50. During the maintenance phase of anesthesia propofol TCI is actively titrated to maintain BIS values between 40 and 50. If BIS is out of this range for more than 10 seconds, propofol is adjusted in 0.5 ug/mc to maintain BIS values in the predetermined limits.
Procedure: Placement of arterial line — An arterial line was placed in the anesthetised patient´s right arm by the investigator and arterial samples were obtained every 10 minutes since initiation of the study infusion to determine plasmatic lidocaine and propofol levels (if the infusion was saline the samples were not analyzed). The arterial line was removed before the end of surgery.

SUMMARY:
The purpose of this randomized clinical trial is to evaluate the interaction of lidocaine infusion initiated and maintained during surgery, on propofol requirements during general anesthesia.

DETAILED DESCRIPTION:
Use of intravenous lidocaine as a coadjuvant agent during general anesthesia has increased. Lidocaine infusion during and after abdominal surgery decreases postoperative pain and reduces ileus duration, reducing patient´s hospital stay and opioid consumption. Intravenous lidocaine´s effect on other intravenous anesthetics is unclear, and there are no present studies evaluating its interaction on hypnotic anesthetic requirements when using a BIS (Bispectral Index) monitor to maintain an adequate depth of anesthesia. We therefore decided to conduct a randomized controlled trial to evaluate the interaction of systemic lidocaine infusion, initiated and maintained during surgery, on propofol requirements and anesthetic depth as measured by BIS.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients,
* Between 20 and 65 years of age
* Programed for elective laparoscopic cholecystectomy
* Eligible for total intravenous anesthesia with propofol

Exclusion Criteria:

* Unwillingness to participate in the study
* Adverse reactions to the drugs used in the study
* Use of medications that interfere in local anesthetic metabolism
* History of liver disease, kidney failure, hypoalbuminemia, hypocalcemia or hypophosphatemia
* History of drug or alcohol abuse
* Chronic use of benzodiazepines

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Total propofol requirements during bispectral index guided general anesthesia | DAY 1.
  During and after elective laparoscopic cholecystectomy. Patients' anesthetic depth will be monitored during the intra-operative period using a BIS monitor. Patients' follow up considers the immediate post-operative period at the recovery room (PACU), and it will continue until patients' discharge from the hospital (average 3 days postoperatively).

SECONDARY OUTCOMES:
Evaluate effect of intravenous lidocaine infusion on waking time after general anesthesia | DAY 1.
  Immediately after elective laparoscopic cholecystectomy, during PACU stay. Patients' follow up considers the immediate post-operative period at the recovery room (PACU), and it will continue until patients' discharge from the hospital (average 3 days postoperatively).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando R Altermatt, MD, Principal Investigator — Departamento de Anestesiología, Hospital Clínico Pontificia Universidad Católica de Chile
Locations (1):
- Hospital Clínico Pontificia Universidad Católica de Chile, Santiago, RM, Chile